CLINICAL TRIAL: NCT02404259
Title: Pharmacokinetics Study of Tenofovir in HIV-infected Thai Children Using Tenofovir-based Regimen
Brief Title: PK TDF in Thai HIV-infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Khon Kaen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HIV-NAT 131
Record Dates: First submitted 2013-02-07; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: HIV
Keywords: pharmacokinetics; TDF; HIV-infected children; Thai; non-nucleoside reverse transcriptase inhibitor (NNRTI); ritonavir-boosted protease inhibitor (bPI); less than eighteen years old
MeSH Terms: interventions — Tenofovir; efavirenz; Lopinavir; Ritonavir; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-nucleoside reverse transcriptase inhibitor (NNRTI) (Other): Efavirenz
  Interventions: Drug: TDF (Tenofovir); Drug: Efavirenz
- ritonavir-boosted protease inhibitor (Other): lopinavir/ritonavir atazanavir/ritonavir
  Interventions: Drug: TDF (Tenofovir); Drug: lopinavir/ritonavir, atazanavir/ritonavir

INTERVENTIONS:
Drug: TDF (Tenofovir)
Drug: Efavirenz
  Arms: non-nucleoside reverse transcriptase inhibitor (NNRTI)
Drug: lopinavir/ritonavir, atazanavir/ritonavir
  Arms: ritonavir-boosted protease inhibitor

SUMMARY:
This study will assess the pharmacokinetics of TDF in Thai HIV-infected children

DETAILED DESCRIPTION:
HIV-infected children who are currently on TDF-base once daily regimen will be enrolled into this study. PK visit will be performed at least 1 month after changing regimen to once daily regimen. Adherence 3 days before PK study will be confirmed using adherence questionnaire. 100% of adherence is needed for PK study. If there is adherence problem on PK visit, PK study will be deferred to at least 3 days. On PK visit, blood drawn will be performed at 0, 2, 4, 6, 8, 10, 12, 24 hr. after taking ARVs for PK study. Blood drawn for safety evaluation will be drawn at any time-point on the PK visit. There is no study drug in this study. All ARVs that patient taking will be according to patient's requirement, and physician judgment. ARVs dosage will follow the Thai national pediatric guideline. CBC, CD4, viral RNA, viral resistance, ALT, cholesterol, and triglyceride results can be from other visits within 4 weeks window period.

Statistical considerations Sample size calculations. There are no pharmacokinetic data in children. In adults, the mean (SD) AUC following administration of a 300mg Viread tablet in fasting state is 2.29 (0.69) microg.hr/mL. In patients taking lopinavir/ritonavir and atazanavir/ritonavir, the mean AUC of TDF is increased by 32% and 24% respectively. Efavirenz does not change the AUC of TDF. If the weight adjusted dose of TDF in children and adolescents achieves the same AUC as in adults and concomitant dosing with a protease inhibitor increases the TDF AUC by 30% but concomitant dosing with Efavirenz does not change the TDF AUC, then 20 treated with Efavirenz and 20 patients treated on a PI based regimen would provide 90% power to detect this difference at the 5% significance level.

Statistical Analysis.

Primary endpoints Pharmacokinetic parameters will be calculated based on individual plasma concentration vs time data, using noncompartmental methods. Data will be summarized overall and by whether the patient is taking a PI or an EFV-based regimen. Formal statistical comparisons of parameters will be made using ANOVA techniques or non-parametric equivalents as appropriate. Effect sizes and 95% confidence intervals will be given for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

* children between the ages of 8-18 years with documented HIV infection
* currently on TDF once daily regimen
* have signed the informed consent

Exclusion Criteria:

* the child or care taker refuse to participate in the study
* severity of adverse events is more than grade 3 thirty days before participating in the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) (pharmacokinetics of TDF) | 12 months
  pharmacokinetics of TDF in children between the ages of 8-18 years

CONTACTS AND LOCATIONS:
Overall Officials: Thanyawee Puthanakit, MD, Principal Investigator — HIV-NAT and Chulalongkorn University
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)'s website — http://www.hivnat.org